CLINICAL TRIAL: NCT00534638
Title: Evaluation of the Effectiveness of Two Vaccination Strategies Using GlaxoSmithKline Biologicals' HPV Vaccine GSK580299 (Cervarix) Administered in Healthy Adolescents
Brief Title: Effectiveness, Safety and Immunogenicity of GSK Biologicals' HPV Vaccine GSK580299 (Cervarix) Administered in Healthy Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 106636; 2007-001731-55 (EudraCT Number)
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Results first posted 2016-01-26 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-10

CONDITIONS: Infections, Papillomavirus
Keywords: HPV vaccine; Healthy adolescents; Cervical cancer; Safety; Immunogenicity; Cervarix
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — human papillomavirus vaccine, L1 type 16, 18; Engerix-B

ARMS (3):
- Cervarix/Engerix-B A Group (Experimental): The A group includes subjects from communities where 70% of male and female adolescents were to be vaccinated with Cervarix vaccine. To achieve a Cervarix vaccination coverage of 70%, a 9:1 ratio was used to allocate study participants to receive Cervarix vaccine versus control Engerix-B vaccine (meaning 90% of vaccinated subjects were randomized to Cervarix). Finally, subjects from A group were either vaccinated with Cervarix, Engerix-B (control vaccine), or not vaccinated (enrolled control without vaccination). Vaccines were administered intramuscularly in the deltoid region of the non-dominant arm according to a 0, 1, 6-month schedule.
  Interventions: Biological: Cervarix; Biological: Engerix-B
- Cervarix/Engerix-B B Group (Experimental): The B group includes subjects from communities where 70% of female adolescents were to be vaccinated with Cervarix vaccine. To achieve a Cervarix vaccination coverage of 70%, a 9:1 ratio was used to allocate female participants to receive Cervarix vaccine versus control Engerix-B vaccine (meaning 90% of vaccinated females were randomized to Cervarix). In this group, all male adolescents were to be vaccinated with Engerix-B control vaccine. Finally, subjects from B group were either vaccinated with Cervarix (females) or Engerix-B/not vaccinated (males and females). Vaccines were administered intramuscularly in the deltoid region of the non-dominant arm according to a 0, 1, 6-month schedule.
  Interventions: Biological: Cervarix; Biological: Engerix-B
- Engerix-B Group (Active Comparator): In this control group, all adolescents were to be vaccinated with Engerix-B control vaccine. Finally, subjects from this group were either vaccinated with Engerix-B or not vaccinated. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm according to a 0, 1, 6-month schedule.
  Interventions: Biological: Engerix-B

INTERVENTIONS:
Biological: Cervarix — Intramuscular injection, 3 doses
  Arms: Cervarix/Engerix-B A Group; Cervarix/Engerix-B B Group
Biological: Engerix-B — Intramuscular injection, 3 doses

SUMMARY:
Genital infections with oncogenic human papillomaviruses (HPV) are common in both men and women. The most important disease associated with oncogenic HPV infection is cervical cancer, currently the second leading cause of cancer-related death among women globally. The current study is designed to evaluate the overall impact of HPV immunization in adolescents 12-15 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Study participants who the investigator or delegate believes that they and/or their parents/legally acceptable representative can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits) should be enrolled in the study.
* A male or female between, and including, 12 and 15 years of age at the time of the first vaccination.

A written informed assent must be obtained from all study participants prior to enrolment. In addition, a written informed consent must be obtained from the study participants' parent or legally acceptable representative.

Note: As according to the Finnish law legal age of consent is 15 years, a written informed consent form can be obtained from study participants aged 15 years old and their parent(s)/legally acceptable representative(s) will receive a letter informing them of their child participation to the study.

* Healthy male and female study participants as established by medical history before entering into the study. If needed, a history-directed clinical examination will be performed by the investigator or delegate (e.g. study nurse).
* Study participants must not be pregnant. Absence of pregnancy should be verified (e.g. urine pregnancy test) as per investigator's or delegate's clinical judgement.
* If the study participant is female, she must be of non-childbearing potential, i.e. be abstinent, have a current tubal ligation, hysterectomy, ovariectomy or be post-menopausal or pre-menarcheal, or if she is of childbearing potential, she must use adequate contraception for 30 days prior to vaccination and continue for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Previous vaccination against HPV or Hepatitis B virus.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* Acute disease at the time of enrolment. (Acute disease is defined as the presence of a moderate or severe illness with or without fever. All vaccines can be administered to persons with a minor illness such as diarrhoea, mild upper respiratory infection with or without low-grade febrile illness, i.e. Oral temperature <37.5°C (99.5°F) / Axillary temperature <37.5°C (99.5°F) / Rectal temperature <38°C (100.4°F).)
* Pregnant or lactating female.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34412 (Actual)
Dates: Start 2007-10-04 (Actual); Primary Completion 2014-12-17 (Actual); Study Completion 2014-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Finland (6):
  - GSK Investigational Site, Kotka
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Rauma
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below).
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=4582

REFERENCES:
- [Background] Lehtinen M, Eriksson T, Apter D, Hokkanen M, Natunen K, Paavonen J, Pukkala E, Angelo MG, Zima J, David MP, Datta S, Bi D, Struyf F, Dubin G. Safety of the human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine in adolescents aged 12-15 years: Interim analysis of a large community-randomized controlled trial. Hum Vaccin Immunother. 2016 Dec;12(12):3177-3185. doi: 10.1080/21645515.2016.1183847. PMID 27841725
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] Adhikari I, Eriksson T, Harjula K, Hokkanen M, Apter D, Nieminen P, Luostarinen T, Lehtinen M. Association of Chlamydia trachomatis infection with cervical atypia in adolescent women with short-term or long-term use of oral contraceptives: a longitudinal study in HPV vaccinated women. BMJ Open. 2022 Jun 1;12(6):e056824. doi: 10.1136/bmjopen-2021-056824. PMID 35649600
- [Derived] Gray P, Kann H, Pimenoff VN, Eriksson T, Luostarinen T, Vanska S, Surcel HM, Faust H, Dillner J, Lehtinen M. Human papillomavirus seroprevalence in pregnant women following gender-neutral and girls-only vaccination programs in Finland: A cross-sectional cohort analysis following a cluster randomized trial. PLoS Med. 2021 Jun 7;18(6):e1003588. doi: 10.1371/journal.pmed.1003588. eCollection 2021 Jun. PMID 34097688
- [Derived] Kalliala I, Eriksson T, Aro K, Hokkanen M, Lehtinen M, Gissler M, Nieminen P. Preterm birth rate after bivalent HPV vaccination: Registry-based follow-up of a randomized clinical trial. Prev Med. 2021 May;146:106473. doi: 10.1016/j.ypmed.2021.106473. Epub 2021 Feb 24. PMID 33639181
- [Derived] Gray P, Kann H, Pimenoff VN, Adhikari I, Eriksson T, Surcel HM, Vanska S, Dillner J, Faust H, Lehtinen M. Long-term follow-up of human papillomavirus type replacement among young pregnant Finnish females before and after a community-randomised HPV vaccination trial with moderate coverage. Int J Cancer. 2020 Dec 15;147(12):3511-3522. doi: 10.1002/ijc.33169. Epub 2020 Jul 7. PMID 32574384
- [Derived] Vanska S, Luostarinen T, Baussano I, Apter D, Eriksson T, Natunen K, Nieminen P, Paavonen J, Pimenoff VN, Pukkala E, Soderlund-Strand A, Dubin G, Garnett G, Dillner J, Lehtinen M. Vaccination With Moderate Coverage Eradicates Oncogenic Human Papillomaviruses If a Gender-Neutral Strategy Is Applied. J Infect Dis. 2020 Aug 17;222(6):948-956. doi: 10.1093/infdis/jiaa099. PMID 32161969
- [Derived] Bi D, Apter D, Eriksson T, Hokkanen M, Zima J, Damaso S, Soila M, Dubin G, Lehtinen M, Struyf F. Safety of the AS04-adjuvanted human papillomavirus (HPV)-16/18 vaccine in adolescents aged 12-15 years: end-of-study results from a community-randomized study up to 6.5 years. Hum Vaccin Immunother. 2020 Jun 2;16(6):1392-1403. doi: 10.1080/21645515.2019.1692557. Epub 2019 Dec 12. PMID 31829767
- [Derived] Lehtinen M, Apter D, Eriksson T, Harjula K, Hokkanen M, Lehtinen T, Natunen K, Damaso S, Soila M, Bi D, Struyf F. Effectiveness of the AS04-adjuvanted HPV-16/18 vaccine in reducing oropharyngeal HPV infections in young females-Results from a community-randomized trial. Int J Cancer. 2020 Jul 1;147(1):170-174. doi: 10.1002/ijc.32791. Epub 2019 Dec 14. PMID 31736068
- [Derived] Lehtinen M, Luostarinen T, Vanska S, Soderlund-Strand A, Eriksson T, Natunen K, Apter D, Baussano I, Harjula K, Hokkanen M, Kuortti M, Palmroth J, Petaja T, Pukkala E, Rekonen S, Siitari-Mattila M, Surcel HM, Tuomivaara L, Paavonen J, Nieminen P, Dillner J, Dubin G, Garnett G. Gender-neutral vaccination provides improved control of human papillomavirus types 18/31/33/35 through herd immunity: Results of a community randomized trial (III). Int J Cancer. 2018 Nov 1;143(9):2299-2310. doi: 10.1002/ijc.31618. Epub 2018 Aug 10. PMID 29845626
- [Derived] Lehtinen M, Soderlund-Strand A, Vanska S, Luostarinen T, Eriksson T, Natunen K, Apter D, Baussano I, Harjula K, Hokkanen M, Kuortti M, Palmroth J, Petaja T, Pukkala E, Rekonen S, Siitari-Mattila M, Surcel HM, Tuomivaara L, Paavonen J, Dillner J, Dubin G, Garnett G. Impact of gender-neutral or girls-only vaccination against human papillomavirus-Results of a community-randomized clinical trial (I). Int J Cancer. 2018 Mar 1;142(5):949-958. doi: 10.1002/ijc.31119. Epub 2017 Nov 9. PMID 29055031
- [Derived] Lehtinen M, Apter D, Baussano I, Eriksson T, Natunen K, Paavonen J, Vanska S, Bi D, David MP, Datta S, Struyf F, Jenkins D, Pukkala E, Garnett G, Dubin G. Characteristics of a cluster-randomized phase IV human papillomavirus vaccination effectiveness trial. Vaccine. 2015 Mar 3;33(10):1284-90. doi: 10.1016/j.vaccine.2014.12.019. Epub 2015 Jan 12. PMID 25593103
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 106636 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106636 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106636 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106636 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106636 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106636 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 106636 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Immunization phase (Day 0 to Month 12) = adolescents (birth cohorts '92-'95) were vaccinated with Cervarix/Engerix-B. Effectiveness evaluation phase (Visit 5) = the vaccine's impact was assessed on female subjects aged 18.5. At Day 0, Cervarix was not licensed for males;male subjects receiving the vaccine were considered part of a Phase III trial.
Pre-assignment Details: 34412 subjects were enrolled in the study, out of which 2236 subjects had a subject number allocated, but did not receive a vaccine dose, and 1 subject was excluded due to non-eligibility criteria, hence 32175 subjects were vaccinated and started the study.
Groups:
- Cervarix Pooled Group: Male and female subjects vaccinated with Cervarix vaccine. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm according to a 0, 1, 6-month schedule.
- Engerix-B Pooled Group: Male and female subjects vaccinated with Engerix-B vaccine. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm according to a 0, 1, 6-month schedule.
Period: Overall Study
Arm/Group | Cervarix Pooled Group | Engerix-B Pooled Group
Started | 14837 | 17338
Completed | 8346 | 5547
Not Completed | 6491 | 11791
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Migrated/moved from study area | 13 | 11
Not completed — Lost to follow-up,incomplete vaccination | 83 | 117
Not completed — Lost to follow-up, complete vaccination | 4707 | 10757
Not completed — Other | 1685 | 902

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix Pooled Group | Engerix-B Pooled Group | Total
Number analyzed (Participants) | 14837 | 17338 | 32175
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.1 (0.8) | 14.1 (0.8) | 14.1 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants] — After the database freeze, discrepancies in the gender of 10 subjects were detected, this leading to 12401 female and 2436 male subjects in the Cervarix Pooled Group, and 8111 female and 9227 male subjects in the Engerix-B Pooled Group.
  These 10 subjects were not part of the Immunogenicity subset, the Diary Card subset or included in the active safety follow-up up to Month 12 for SAEs.
  These 10 subjects did not report any AEs and did not have any sample results. The impact on the AEs and overall effectiveness analysis was limited to the number of subjects exposed and considered minor.
  Participants
    Female | 12399 | 8119 | 20518
    Male | 2438 | 9219 | 11657
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African heritage/African American | 9 | 8 | 17
  Geographic ancestry: Asian - Central/South Asian heritage | 3 | 4 | 7
  Geographic ancestry: Asian - East Asian heritage | 8 | 0 | 8
  Geographic ancestry: Asian - Japanese heritage | 1 | 1 | 2
  Geographic ancestry: Asian - South East Asian heritage | 13 | 4 | 17
  Geographic ancestry: White - Arabic/North African heritage | 31 | 39 | 70
  Geographic ancestry: White - Caucasian/European heritage | 14669 | 17190 | 31859
  Geographic ancestry: Mixed origin | 103 | 92 | 195

OUTCOME MEASURES:

1. Primary Outcome: Number of Female Subjects With Overall Vaccine Effectiveness Against Genital Infection With Human Papilloma Virus (HPV)-16/18 Types in Cervarix/Engerix-B B Group Versus Engerix-B Group and in Cervarix/Engerix-B A Group Versus Engerix-B Group
Description: The analysis of overall effectiveness of Cervarix vaccine against genital infection with HPV-16/18 types was based on stratified Mantel-Haenszel adjusted for clustering. The overall vaccine effectiveness was computed as 1- the prevalence odd ratio in all subjects from the investigated group (prevalence rate in all subjects from the investigated group/prevalence rate in all subjects from Engerix-B Group).
Time Frame: At the time of Visit 5 (i.e. at 18.5 years of age)
Population: The analysis was performed on female study participants from the Total Enrolled cohort on effectiveness, which included all study participants who were previously enrolled in the immunization phase, and those who joined the trial at Visit 5, for whom results were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix/Engerix-B A Group | Cervarix/Engerix-B B Group | Engerix-B Group
Number analyzed (Participants) | 3629 | 4029 | 3168
Participants | 139 | 117 | 329
Statistical Analysis 1: Comparison: Cervarix/Engerix-B B Group vs Engerix-B Group; Overall efectiveness against HPV-16/18 Cervarix/Engerix-B B Group vs Engerix-B Group: The analysis of the overall effectiveness of GSK's HPV-16/18 vaccine against HPV-16/18 genital infection in Cervarix/Engerix-B B Group versus Engerix-B Group was based on stratified Mantel-Haenszel adjusted for clustering; Test type: Superiority; p = 0.004, Cochran-Mantel-Haenszel — An objective was reached if the 2-sided p-value associated to the objective was below 5%; Vaccine effectiveness percentage = 49.6, 95% CI 2-sided [20.1 to 68.2]
Statistical Analysis 2: Comparison: Cervarix/Engerix-B A Group vs Engerix-B Group; Overall efectiveness against HPV-16/18 Cervarix/Engerix-B A Group vs Engerix-B Group: The analysis of the overall effectiveness of GSK's HPV-16/18 vaccine against HPV-16/18 genital infection in Cervarix/Engerix-B A Group versus Engerix-B Group was based on stratified Mantel-Haenszel adjusted for clustering; Test type: Superiority; p = 0.232, Cochran-Mantel-Haenszel — An objective was reached if the 2-sided p-value associated to the objective was below 5%; Vaccine effectiveness percentage = 23.8, 95% CI 2-sided [-19.0 to 51.1]

2. Secondary Outcome: Number of Female Subjects With Overall Vaccine Effectiveness Against Genital Infection With HPV-16/18 Types in Cervarix/Engerix-B A Group Versus Cervarix/Engerix-B B Group
Description: The analysis of overall effectiveness of Cervarix vaccine against genital infection with HPV-16/18 types was based on stratified Mantel-Haenszel adjusted for clustering. The overall vaccine effectiveness was computed as 1- the prevalence odd ratio in all subjects from the investigated group (prevalence rate in all subjects from the Cervarix/Engerix-B A Group/prevalence rate in all subjects from Engerix-B Group).
  Note: As per Protocol and as the confirmatory objectives were not met, only exploratory interpretation could be performed for what concerns this secondary outcome measure.
Time Frame: At the time of Visit 5 (i.e. at 18.5 years of age)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix/Engerix-B A Group | Cervarix/Engerix-B B Group
Number analyzed (Participants) | 3629 | 4029
Participants | 139 | 117
Statistical Analysis 1: Comparison: Cervarix/Engerix-B A Group vs Cervarix/Engerix-B B Group; Overall efectiveness against HPV-16/18 Cervarix/Engerix-B A Group vs Cervarix/Engerix-B B Group: The analysis of the overall effectiveness of GSK's HPV-16/18 vaccine against HPV-16/18 genital infection in Cervarix/Engerix-B A Group versus Cervarix/Engerix-B B was based on stratified Mantel-Haenszel adjusted for clustering; Test type: Superiority; p = 0.069, Cochran-Mantel-Haenszel — An objective was reached if the 2-sided p-value associated to the objective was below 5%; Vaccine effectiveness percentage = -52.2, 95% CI 2-sided [-139.4 to 3.3]

3. Secondary Outcome: Number of Female Subjects With Overall Vaccine Effectiveness Against Genital Oncogenic Infection With Specific HPV Types
Description: The analysis of overall effectiveness of Cervarix vaccine against genital infection with specific HPV types (16, 18, 31/45, 31/33/45, 31/33/45/51, 31/33/45/51/52, 31/33/35/39/45/51/52/56/58/59/66/68, 16/18/31/33/35/39/45/51/52/56/58/59/66/68, 6, 11, 6/11, 6/11/53/74) was based on stratified Mantel-Haenszel adjusted for clustering. The effectiveness was computed as 1- the prevalence odd ratio in all subjects from the investigated group (prevalence rate in all subjects from the investigated group/prevalence rate in all subjects from Engerix-B Group).
Time Frame: At the time of Visit 5 (i.e. at 18.5 years of age)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix/Engerix-B A Group | Cervarix/Engerix-B B Group | Engerix-B Group
Number analyzed (Participants) | 3629 | 4029 | 3168
Participants
  HPV-16 | 88 | 85 | 227
  HPV-18 | 62 | 41 | 134
  HPV-31/45 | 97 | 93 | 182
  HPV-31/33/45 | 175 | 173 | 271
  HPV-31/33/45/51 | 449 | 450 | 441
  HPV-31/33/45/51/52 | 563 | 585 | 532
  HPV-31/33/35/39/45/51/52/56/58/59/66/68 | 923 | 961 | 776
  HPV-16/18/31/33/35/39/45/51/52/56/58/59/66/68 | 965 | 999 | 883
  HPV-6 | 192 | 183 | 139
  HPV-11 | 39 | 32 | 34
  HPV-6/11 | 221 | 204 | 165
  HPV-6/11/53/74 | 403 | 381 | 307

4. Secondary Outcome: Number of Female Subjects With Total Vaccine Effectiveness Against Oropharyngeal Infection With HPV-16/18 Types
Description: The analysis of total effectiveness of Cervarix vaccine against oropharyngeal infection with HPV-16/18 types was based on stratified Mantel-Haenszel adjusted for clustering. The effectiveness was computed as 1- the prevalence odd ratio in Cervarix vaccinated subjects from the investigated group (prevalence rate in Cervarix vaccinated subjects from the investigated group/prevalence rate in all subjects from Engerix-B Group).
Time Frame: At the time of Visit 5 (i.e. at 18.5 years of age)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Cervarix/Engerix-B Pooled Group: Pooled A and B group: This pooled group includes subjects from communities where 70% of male and female adolescents (A group) or 70% of female adolescents (B group) were to be vaccinated with Cervarix vaccine. To achieve a Cervarix vaccination coverage of 70%, a 9:1 ratio was used to allocate study participants (A group) or female participants (B group) to receive Cervarix vaccine versus control Engerix-B vaccine (meaning 90% of vaccinated subjects (A group) or vaccinated females (B group) were randomized to Cervarix). Finally, subjects from this pooled group were either vaccinated with Cervarix, Engerix-B (control vaccine), or not vaccinated (enrolled control without vaccination). Vaccines were administered intramuscularly in the deltoid region of the non-dominant arm according to a 0, 1, 6-month schedule.
Arm/Group | Cervarix/Engerix-B Pooled Group | Engerix-B Group
Number analyzed (Participants) | 3192 | 1679
Participants | 9 | 27

5. Secondary Outcome: Number of Female Subjects With Total Vaccine Effectiveness Against Oropharyngeal Oncogenic Infection With Specific HPV Types
Description: The analysis of total effectiveness of Cervarix vaccine against oropharyngeal infection with specific HPV types (16, 18, 31/45, 31/33/45, 31/33/45/51, 31/33/45/51/52, 31/33/35/39/45/51/52/56/58/59/66/68, 16/18/31/33/35/39/45/51/52/56/58/59/66/68, 6, 11, 6/11, 6/11/53/74) was based on stratified Mantel-Haenszel adjusted for clustering. The effectiveness was computed as 1- the prevalence odd ratio in all Cervarix vaccinated subjects from the investigated group (prevalence rate in all Cervarix vaccinated subjects from the investigated group/prevalence rate in all subjects from Engerix-B Group).
Time Frame: At the time of Visit 5 (at 18.5 years of age)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix/Engerix-B Pooled Group | Engerix-B Group
Number analyzed (Participants) | 3192 | 1679
Participants
  HPV-16 | 6 | 19
  HPV-18 | 4 | 10
  HPV-31/45 | 3 | 9
  HPV-31/33/45 | 9 | 16
  HPV-31/33/45/51 | 53 | 42
  HPV-31/33/45/51/52 | 63 | 49
  HPV-31/33/35/39/45/51/52/56/58/59/66/68 | 129 | 79
  HPV-16/18/31/33/35/39/45/51/52/56/58/59/66/68 | 136 | 95
  HPV-6 | 36 | 27
  HPV-11 | 5 | 5
  HPV-6/11 | 41 | 29
  HPV-6/11/53/74 | 72 | 45

6. Secondary Outcome: Number of Male Subjects Reporting Any and Grade 3 Solicited Local Symptoms, in a Subset of Subjects
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 7-day post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total vaccinated cohort (TVC) - the Diary card subset, which included a subset of male adolescents from Cervarix/Engerix-B A Group and Engerix-B Group, with at least one study vaccine administration documented, who were selected for active assessment of safety using diary cards and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Pooled Group | Engerix-B Pooled Group
Number analyzed (Participants) | 603 | 1028
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 590 | 1021
  Any Pain, Dose 1 | 463 | 157
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 590 | 1021
  Grade 3 Pain, Dose 1 | 12 | 1
  Any Redness, Dose 1: number analyzed (Participants) | 590 | 1021
  Any Redness, Dose 1 | 99 | 90
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 590 | 1021
  Grade 3 Redness, Dose 1 | 1 | 0
  Any Swelling, Dose 1: number analyzed (Participants) | 590 | 1021
  Any Swelling, Dose 1 | 61 | 29
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 590 | 1021
  Grade 3 Swelling, Dose 1 | 4 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 509 | 935
  Any Pain, Dose 2 | 331 | 123
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 509 | 935
  Grade 3 Pain, Dose 2 | 9 | 1
  Any Redness, Dose 2: number analyzed (Participants) | 509 | 935
  Any Redness, Dose 2 | 88 | 59
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 509 | 935
  Grade 3 Redness, Dose 2 | 1 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 509 | 935
  Any Swelling, Dose 2 | 66 | 16
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 509 | 935
  Grade 3 Swelling, Dose 2 | 3 | 0
  Any Pain, Dose 3: number analyzed (Participants) | 491 | 812
  Any Pain, Dose 3 | 326 | 108
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 491 | 812
  Grade 3 Pain, Dose 3 | 11 | 0
  Any Redness, Dose 3: number analyzed (Participants) | 491 | 812
  Any Redness, Dose 3 | 100 | 50
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 491 | 812
  Grade 3 Redness, Dose 3 | 2 | 0
  Any Swelling, Dose 3: number analyzed (Participants) | 491 | 812
  Any Swelling, Dose 3 | 69 | 18
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 491 | 812
  Grade 3 Swelling, Dose 3 | 3 | 0
  Any Pain, Across doses | 506 | 251
  Grade 3 Pain, Across doses | 26 | 2
  Any Redness, Across doses | 169 | 131
  Grade 3 Redness, Across doses | 4 | 0
  Any Swelling, Across doses | 131 | 46
  Grade 3 Swelling, Across doses | 8 | 0

7. Secondary Outcome: Number of Male Subjects Reporting Any, Grade 3 and Related to Vaccination Solicited General Symptoms, in a Subset of Subjects
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], gastrointestinal symptoms (including nausea, vomiting, diarrhoea and/or abdominal pain), headache, myalgia, rash and urticaria. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day post-vaccination period following each dose and across doses
Population: The analysis was performed on the TVC - the Diary card subset, which included a subset of male adolescents from Cervarix/Engerix-B A Group and Engerix-B Group, with at least one study vaccine administration documented, who were selected for active assessment of safety using diary cards and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Pooled Group | Engerix-B Pooled Group
Number analyzed (Participants) | 604 | 1028
Participants
  Any Arthralgia, Dose 1: number analyzed (Participants) | 590 | 1021
  Any Arthralgia, Dose 1 | 58 | 58
  Grade 3 Arthralgia, Dose 1: number analyzed (Participants) | 590 | 1021
  Grade 3 Arthralgia, Dose 1 | 0 | 1
  Related Arthralgia, Dose 1: number analyzed (Participants) | 590 | 1021
  Related Arthralgia, Dose 1 | 37 | 45
  Any Fatigue, Dose 1: number analyzed (Participants) | 590 | 1021
  Any Fatigue, Dose 1 | 224 | 301
  Grade 3 Fatigue, Dose 1: number analyzed (Participants) | 590 | 1021
  Grade 3 Fatigue, Dose 1 | 3 | 9
  Related Fatigue, Dose 1: number analyzed (Participants) | 590 | 1021
  Related Fatigue, Dose 1 | 156 | 246
  Any Fever (axillary), Dose 1: number analyzed (Participants) | 590 | 1021
  Any Fever (axillary), Dose 1 | 15 | 35
  Grade 3 Fever (axillary), Dose 1: number analyzed (Participants) | 590 | 1021
  Grade 3 Fever (axillary), Dose 1 | 3 | 4
  Related Fever (axillary), Dose 1: number analyzed (Participants) | 590 | 1021
  Related Fever (axillary), Dose 1 | 7 | 23
  Any Gastrointestinal, Dose 1: number analyzed (Participants) | 590 | 1021
  Any Gastrointestinal, Dose 1 | 73 | 101
  Grade 3 Gastrointestinal, Dose 1: number analyzed (Participants) | 590 | 1021
  Grade 3 Gastrointestinal, Dose 1 | 7 | 6
  Related Gastrointestinal, Dose 1: number analyzed (Participants) | 590 | 1021
  Related Gastrointestinal, Dose 1 | 45 | 84
  Any Headache, Dose 1: number analyzed (Participants) | 590 | 1021
  Any Headache, Dose 1 | 178 | 255
  Grade 3 Headache, Dose 1: number analyzed (Participants) | 590 | 1021
  Grade 3 Headache, Dose 1 | 10 | 7
  Related Headache, Dose 1: number analyzed (Participants) | 590 | 1021
  Related Headache, Dose 1 | 108 | 181
  Any Myalgia, Dose 1: number analyzed (Participants) | 590 | 1021
  Any Myalgia, Dose 1 | 229 | 169
  Grade 3 Myalgia, Dose 1: number analyzed (Participants) | 590 | 1021
  Grade 3 Myalgia, Dose 1 | 6 | 2
  Related Myalgia, Dose 1: number analyzed (Participants) | 590 | 1021
  Related Myalgia, Dose 1 | 196 | 138
  Any Rash, Dose 1: number analyzed (Participants) | 590 | 1021
  Any Rash, Dose 1 | 13 | 17
  Grade 3 Rash, Dose 1: number analyzed (Participants) | 590 | 1021
  Grade 3 Rash, Dose 1 | 0 | 0
  Related Rash, Dose 1: number analyzed (Participants) | 590 | 1021
  Related Rash, Dose 1 | 5 | 12
  Any Urticaria, Dose 1: number analyzed (Participants) | 590 | 1021
  Any Urticaria, Dose 1 | 3 | 12
  Grade 3 Urticaria, Dose 1: number analyzed (Participants) | 590 | 1021
  Grade 3 Urticaria, Dose 1 | 0 | 0
  Related Urticaria, Dose 1: number analyzed (Participants) | 590 | 1021
  Related Urticaria, Dose 1 | 2 | 11
  Any Arthralgia, Dose 2: number analyzed (Participants) | 511 | 936
  Any Arthralgia, Dose 2 | 41 | 38
  Grade 3 Arthralgia, Dose 2: number analyzed (Participants) | 511 | 936
  Grade 3 Arthralgia, Dose 2 | 0 | 3
  Related Arthralgia, Dose 2: number analyzed (Participants) | 511 | 936
  Related Arthralgia, Dose 2 | 36 | 33
  Any Fatigue, Dose 2: number analyzed (Participants) | 511 | 936
  Any Fatigue, Dose 2 | 136 | 155
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 511 | 936
  Grade 3 Fatigue, Dose 2 | 2 | 7
  Related Fatigue, Dose 2: number analyzed (Participants) | 511 | 936
  Related Fatigue, Dose 2 | 100 | 123
  Any Fever, Dose 2: number analyzed (Participants) | 511 | 936
  Any Fever, Dose 2 | 19 | 28
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 511 | 936
  Grade 3 Fever, Dose 2 | 1 | 2
  Related Fever, Dose 2: number analyzed (Participants) | 511 | 936
  Related Fever, Dose 2 | 11 | 10
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 511 | 936
  Any Gastrointestinal, Dose 2 | 45 | 50
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 511 | 936
  Grade 3 Gastrointestinal, Dose 2 | 4 | 5
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 511 | 936
  Related Gastrointestinal, Dose 2 | 27 | 38
  Any Headache, Dose 2: number analyzed (Participants) | 511 | 936
  Any Headache, Dose 2 | 101 | 144
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 511 | 936
  Grade 3 Headache, Dose 2 | 5 | 4
  Related Headache, Dose 2: number analyzed (Participants) | 511 | 936
  Related Headache, Dose 2 | 55 | 104
  Any Myalgia, Dose 2: number analyzed (Participants) | 511 | 936
  Any Myalgia, Dose 2 | 151 | 97
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 511 | 936
  Grade 3 Myalgia, Dose 2 | 1 | 1
  Related Myalgia, Dose 2: number analyzed (Participants) | 511 | 936
  Related Myalgia, Dose 2 | 143 | 77
  Any Rash, Dose 2: number analyzed (Participants) | 511 | 936
  Any Rash, Dose 2 | 9 | 14
  Grade 3 Rash, Dose 2: number analyzed (Participants) | 511 | 936
  Grade 3 Rash, Dose 2 | 0 | 0
  Related Rash, Dose 2: number analyzed (Participants) | 511 | 936
  Related Rash, Dose 2 | 4 | 9
  Any Urticaria, Dose 2: number analyzed (Participants) | 511 | 936
  Any Urticaria, Dose 2 | 1 | 2
  Grade 3 Urticaria, Dose 2: number analyzed (Participants) | 511 | 936
  Grade 3 Urticaria, Dose 2 | 0 | 0
  Related Urticaria, Dose 2: number analyzed (Participants) | 511 | 936
  Related Urticaria, Dose 2 | 1 | 1
  Any Arthralgia, Dose 3: number analyzed (Participants) | 492 | 814
  Any Arthralgia, Dose 3 | 53 | 33
  Grade 3 Arthralgia, Dose 3: number analyzed (Participants) | 492 | 814
  Grade 3 Arthralgia, Dose 3 | 1 | 0
  Related Arthralgia, Dose 3: number analyzed (Participants) | 492 | 814
  Related Arthralgia, Dose 3 | 41 | 29
  Any Fatigue, Dose 3: number analyzed (Participants) | 492 | 814
  Any Fatigue, Dose 3 | 135 | 141
  Grade 3 Fatigue, Dose 3: number analyzed (Participants) | 492 | 814
  Grade 3 Fatigue, Dose 3 | 4 | 6
  Related Fatigue, Dose 3: number analyzed (Participants) | 492 | 814
  Related Fatigue, Dose 3 | 100 | 116
  Any Fever, Dose 3: number analyzed (Participants) | 492 | 814
  Any Fever, Dose 3 | 15 | 27
  Grade 3 Fever, Dose 3: number analyzed (Participants) | 492 | 814
  Grade 3 Fever, Dose 3 | 2 | 3
  Related Fever, Dose 3: number analyzed (Participants) | 492 | 814
  Related Fever, Dose 3 | 10 | 24
  Any Gastrointestinal, Dose 3: number analyzed (Participants) | 492 | 814
  Any Gastrointestinal, Dose 3 | 19 | 50
  Grade 3 Gastrointestinal, Dose 3: number analyzed (Participants) | 492 | 814
  Grade 3 Gastrointestinal, Dose 3 | 0 | 2
  Related Gastrointestinal, Dose 3: number analyzed (Participants) | 492 | 814
  Related Gastrointestinal, Dose 3 | 12 | 39
  Any Headache, Dose 3: number analyzed (Participants) | 492 | 814
  Any Headache, Dose 3 | 101 | 123
  Grade 3 Headache, Dose 3: number analyzed (Participants) | 492 | 814
  Grade 3 Headache, Dose 3 | 2 | 3
  Related Headache, Dose 3: number analyzed (Participants) | 492 | 814
  Related Headache, Dose 3 | 69 | 97
  Any Myalgia, Dose 3: number analyzed (Participants) | 492 | 814
  Any Myalgia, Dose 3 | 158 | 80
  Grade 3 Myalgia, Dose 3: number analyzed (Participants) | 492 | 814
  Grade 3 Myalgia, Dose 3 | 5 | 0
  Related Myalgia, Dose 3: number analyzed (Participants) | 492 | 814
  Related Myalgia, Dose 3 | 137 | 69
  Any Rash, Dose 3: number analyzed (Participants) | 492 | 814
  Any Rash, Dose 3 | 11 | 9
  Grade 3 Rash, Dose 3: number analyzed (Participants) | 492 | 814
  Grade 3 Rash, Dose 3 | 0 | 0
  Related Rash, Dose 3: number analyzed (Participants) | 492 | 814
  Related Rash, Dose 3 | 5 | 8
  Any Urticaria, Dose 3: number analyzed (Participants) | 492 | 814
  Any Urticaria, Dose 3 | 0 | 3
  Grade 3 Urticaria, Dose 3: number analyzed (Participants) | 492 | 814
  Grade 3 Urticaria, Dose 3 | 0 | 0
  Related Urticaria, Dose 3: number analyzed (Participants) | 492 | 814
  Related Urticaria, Dose 3 | 0 | 3
  Any Arthralgia, Across doses | 107 | 97
  Grade 3 Arthralgia, Across doses | 1 | 4
  Related Arthralgia, Across doses | 87 | 81
  Any Fatigue, Across doses | 291 | 411
  Grade 3 Fatigue, Across doses | 7 | 21
  Related Fatigue, Across doses | 233 | 351
  Any Fever, Across doses | 48 | 85
  Grade 3 Fever, Across doses | 6 | 9
  Related Fever, Across doses | 28 | 53
  Any Gastrointestinal, Across doses | 106 | 163
  Grade 3 Gastrointestinal, Across doses | 11 | 13
  Related Gastrointestinal, Across doses | 70 | 128
  Any Headache, Across doses | 261 | 371
  Grade 3 Headache, Across doses | 15 | 14
  Related Headache, Across doses | 176 | 280
  Any Myalgia, Across doses | 321 | 250
  Grade 3 Myalgia, Across doses | 12 | 3
  Related Myalgia, Across doses | 291 | 211
  Any Rash, Across doses | 29 | 33
  Grade 3 Rash, Across doses | 0 | 0
  Related Rash, Across doses | 14 | 23
  Any Urticaria, Across doses | 4 | 15
  Grade 3 Urticaria, Across doses | 0 | 0
  Related Urticaria, Across doses | 3 | 13

8. Secondary Outcome: Number of Male Subjects Reporting Any, Grade 3 and Related to Vaccination Unsolicited Adverse Events (AEs), in a Subset of Subjects
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within the 30-day post-vaccination period
Population: This analysis was performed on the TVC - the Diary Card subset, which included a subset of male adolescents from Cervarix/Engerix-B A Group and Engerix-B Group who were selected for active assessment of safety using diary cards and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Pooled Group | Engerix-B Pooled Group
Number analyzed (Participants) | 643 | 1047
Participants
  Any AEs | 157 | 202
  Grade 3 AEs | 31 | 46
  Related AEs | 12 | 19

9. Secondary Outcome: Number of Male Subjects With Urticaria/Rash Within 30 Minutes After Each Vaccination Dose, in a Subset of Subjects
Description: The number of subjects with urticaria/rash assessed within 30 minutes following each vaccine dose are reported. Confirmed urticaria/rash = subjects who reported urticaria/rash within the specified time frame. Not confirmed urticaria/rash = number of subjects who did not report urticaria/rash within the specified time frame.
Time Frame: Within 30 minutes following each vaccination dose
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Pooled Group | Engerix-B Pooled Group
Number analyzed (Participants) | 643 | 1047
Participants
  Not confirmed urticaria/rash, Dose 1 | 643 | 1047
  Confirmed urticaria/rash, Dose 1 | 0 | 0
  Not confirmed urticaria/rash, Dose 2: number analyzed (Participants) | 634 | 1042
  Not confirmed urticaria/rash, Dose 2 | 634 | 1042
  Confirmed urticaria/rash, Dose 2: number analyzed (Participants) | 634 | 1042
  Confirmed urticaria/rash, Dose 2 | 0 | 0
  Not confirmed urticaria/rash, Dose 3: number analyzed (Participants) | 631 | 1039
  Not confirmed urticaria/rash, Dose 3 | 630 | 1039
  Confirmed urticaria/rash, Dose 3: number analyzed (Participants) | 631 | 1039
  Confirmed urticaria/rash, Dose 3 | 0 | 0
  Missing urticaria/rash, Dose 3: number analyzed (Participants) | 631 | 1039
  Missing urticaria/rash, Dose 3 | 1 | 0

10. Secondary Outcome: Number of Male Subjects Reporting Medically Significant Conditions (MSCs), in a Subset of Subjects
Description: MSCs are defined as AEs prompting emergency room or physician visits that are not (1) related to common diseases or (2) routine visits for physical examination or vaccination, or SAEs that are not related to common diseases. Common diseases include: upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections and injury.
Time Frame: From Dose 1 (at Day 0) until Month 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Pooled Group | Engerix-B Pooled Group
Number analyzed (Participants) | 643 | 1047
Participants | 47 | 76

11. Secondary Outcome: Number of Male Subjects Reporting Any Serious Adverse Events (SAEs) and SAEs Causally Related to Vaccination, in a Subset of Subjects
Description: Serious adverse events (SAEs) assessed include medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity.
Time Frame: From Dose 1 (at Day 0) until Month 12
Population: The analysis was performed on the TVC - subset of male subjects with active follow-up Month 0-Month 12 for SAEs, which included the male subjects in the Diary Card subset and the remaining Cervarix/Engerix-B A Group male subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Pooled Group | Engerix-B Pooled Group
Number analyzed (Participants) | 2436 | 1267
Participants
  Any SAEs | 58 | 25
  Related SAEs | 4 | 1

12. Secondary Outcome: Number of Subjects Reporting SAEs Assessed by the Investigator as Possibly Related to Vaccination
Description: as for outcome 11
Time Frame: During the entire study period (from Day 0 up to Visit 5 [18.5 years of age] or up to the day before 19 years of age for subjects who did not attend Visit 5)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Pooled Group | Engerix-B Pooled Group
Number analyzed (Participants) | 14837 | 17338
Participants | 25 | 30

13. Secondary Outcome: Number of Subjects With New Onset of Autoimmune Diseases (NOADs), Retrieved From Care Register for Social Welfare and Health Care (HILMO)
Description: NOADs include colitis ulcerative, juvenile arthritis, type 1 diabetes mellitus, coeliac disease and Chron's disease, Basedow's disease, erythema nodosum VIIth nerve paralysis and psoriasis.
Time Frame: During the entire study period (from day 0 up to Visit 5 [at 18.5 years of age] or up to the day before 19 years of age for subjects who did not attend Visit 5)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Pooled Group | Engerix-B Pooled Group
Number analyzed (Participants) | 14837 | 17338
Participants | 149 | 180

14. Secondary Outcome: Number of Subjects Reporting Pregnancies and Outcomes of Reported Pregnancies With Onset During the Study Period, Retrieved From Medical Birth Registry and HILMO
Description: Pregnancies with onset during the study were classified by their outcome. Outcomes included live infant with no apparent congenital anomaly, elective termination with no apparent congenital anomaly, spontaneous abortion with no apparent congenital anomaly, ectopic pregnancy, stillbirth with no apparent congenital anomaly and molar pregnancy.
  Note: The analysis was performed based on the corrected demographical data. Please refer to the rationale provided in the Baseline characteristics section.
Time Frame: as for outcome 13
Population: The analysis was performed on the total number of pregnant subjects reported, part of the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Pooled Group | Engerix-B Pooled Group
Number analyzed (Participants) | 777 | 567
Participants
  Live infant with no apparent anomaly | 254 | 183
  Elective termination with no apparent anomaly | 454 | 332
  Ectopic pregnancy | 5 | 5
  Spontaneous abortion with no apparent anomaly | 62 | 45
  Stillbirth with no apparent congenital anomaly | 0 | 1
  Molar pregnancy | 2 | 1

15. Secondary Outcome: Number of Subjects With HPV-16 and HPV-18 Antibody Concentrations Equal to or Above the Cut-off Values, by Gender, in a Subset of Subjects
Description: The antibody concentrations against HPV-16 and HPV-18 were determined by Enzyme-linked immunosorbent assay (ELISA). The cut-off of the assay was 8 ELISA units per milliliter (EL.U/mL) for anti-HPV-16 and 7 EL.U/mL for anti-HPV-18 at Visits 1 and 4 and 19 EL.U/mL for HPV-16 and 18 EL.U/mL for HPV-18 at Visit 5.
Time Frame: At the time of Visit 1 (at Day 0), Visit 4 (at Month 7) and Visit 5 (at 18.5 years of age)
Population: The analysis was performed on the ATP cohort for immunogenicity-Immunogenicity subset, which comprised the same male study subjects from the Cervarix/Engerix-B A Group included in the Diary Card subset, plus approximately 1500 female study subjects from the same Cervarix/Engerix-B A Group, with assay results available at the considered time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Pooled Group
Number analyzed (Participants) | 1163
Participants
  anti-HPV-16 ≥ 8 EL.U/mL, males (Day 0): number analyzed (Participants) | 536
  anti-HPV-16 ≥ 8 EL.U/mL, males (Day 0) | 40
  anti-HPV-16 ≥ 8 EL.U/mL, males (Month 7): number analyzed (Participants) | 536
  anti-HPV-16 ≥ 8 EL.U/mL, males (Month 7) | 536
  anti-HPV-16 ≥ 19 EL.U/mL, males (18.5Y): number analyzed (Participants) | 217
  anti-HPV-16 ≥ 19 EL.U/mL, males (18.5Y) | 217
  anti-HPV-16 ≥ 8 EL.U/mL, females (Day 0) | 86
  anti-HPV-16 ≥ 8 EL.U/mL, females (Month 7) | 1163
  anti-HPV-16 ≥ 19 EL.U/mL, females (18.5Y): number analyzed (Participants) | 688
  anti-HPV-16 ≥ 19 EL.U/mL, females (18.5Y) | 688
  anti-HPV-18 ≥ 7 EL.U/mL, males (Day 0): number analyzed (Participants) | 535
  anti-HPV-18 ≥ 7 EL.U/mL, males (Day 0) | 31
  anti-HPV-18 ≥ 7 EL.U/mL, males (Month 7): number analyzed (Participants) | 535
  anti-HPV-18 ≥ 7 EL.U/mL, males (Month 7) | 535
  anti-HPV-18 ≥ 18 EL.U/mL, males (18.5Y): number analyzed (Participants) | 217
  anti-HPV-18 ≥ 18 EL.U/mL, males (18.5Y) | 217
  anti-HPV-18 ≥ 7 EL.U/mL, females (Day 0): number analyzed (Participants) | 1160
  anti-HPV-18 ≥ 7 EL.U/mL, females (Day 0) | 84
  anti-HPV-18 ≥ 7 EL.U/mL, females (Month 7): number analyzed (Participants) | 1160
  anti-HPV-18 ≥ 7 EL.U/mL, females (Month 7) | 1160
  anti-HPV-18 ≥ 18 EL.U/mL, females (18.5Y): number analyzed (Participants) | 686
  anti-HPV-18 ≥ 18 EL.U/mL, females (18.5Y) | 685

16. Secondary Outcome: Anti-HPV-16 and Anti-HPV-18 Antibody Concentrations, by Gender, in a Subset of Subjects
Description: as for outcome 15
Time Frame: At the time of Visit 1 (Day 0), Visit 4 (at Month 7) and at the time of Visit 5 (18.5 years of age)
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Pooled Group
Number analyzed (Participants) | 1163
EL.U/mL
  anti-HPV-16 ≥ 8 EL.U/mL, males (Day 0): number analyzed (Participants) | 536
  anti-HPV-16 ≥ 8 EL.U/mL, males (Day 0) | 4.5 [4.3 to 4.6]
  anti-HPV-16 ≥ 8 EL.U/mL, males (Month 7): number analyzed (Participants) | 536
  anti-HPV-16 ≥ 8 EL.U/mL, males (Month 7) | 23959.1 [22301.0 to 25740.4]
  anti-HPV-16 ≥ 19 EL.U/mL, males (18.5Y): number analyzed (Participants) | 217
  anti-HPV-16 ≥ 19 EL.U/mL, males (18.5Y) | 2759.5 [2432.1 to 3130.9]
  anti-HPV-16 ≥ 8 EL.U/mL, females (Day 0) | 4.5 [4.4 to 4.6]
  anti-HPV-16 ≥ 8 EL.U/mL, females (Month 7) | 21327.2 [20338.9 to 22363.5]
  anti-HPV-16 ≥ 19 EL.U/mL, females (18.5Y): number analyzed (Participants) | 688
  anti-HPV-16 ≥ 19 EL.U/mL, females (18.5Y) | 2609.6 [2444.4 to 2785.9]
  anti-HPV-18 ≥ 7 EL.U/mL, males (Day 0): number analyzed (Participants) | 535
  anti-HPV-18 ≥ 7 EL.U/mL, males (Day 0) | 3.8 [3.7 to 4.0]
  anti-HPV-18 ≥ 7 EL.U/mL, males (Month 7): number analyzed (Participants) | 535
  anti-HPV-18 ≥ 7 EL.U/mL, males (Month 7) | 8583.9 [7974.7 to 9239.5]
  anti-HPV-18 ≥ 18 EL.U/mL, males (18.5Y): number analyzed (Participants) | 217
  anti-HPV-18 ≥ 18 EL.U/mL, males (18.5Y) | 837.7 [727.3 to 964.9]
  anti-HPV-18 ≥ 7 EL.U/mL, females (Day 0): number analyzed (Participants) | 1160
  anti-HPV-18 ≥ 7 EL.U/mL, females (Day 0) | 3.9 [3.8 to 4.0]
  anti-HPV-18 ≥ 7 EL.U/mL, females (Month 7): number analyzed (Participants) | 1160
  anti-HPV-18 ≥ 7 EL.U/mL, females (Month 7) | 8227.3 [7847.7 to 8625.4]
  anti-HPV-18 ≥ 18 EL.U/mL, females (18.5Y): number analyzed (Participants) | 686
  anti-HPV-18 ≥ 18 EL.U/mL, females (18.5Y) | 890.0 [826.2 to 958.7]

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during the 7-day post-vaccination period (across doses). Unsolicited AEs: within the 30-day post-vaccination period (across doses). SAEs: during the entire study period (from Day 0 up to Visit 5 [at 18.5 years of age] or up to the day before 19 years of age for subjects who did not attend Visit 5).
Description: AEs were collected in the TVC-Diary Card subset. For this study, the Total Number of Participants Affected by Other (non-serious) AEs was analyzed separately for solicited AEs and for unsolicited AEs. A consolidated analysis of all solicited and unsolicited AEs was not technically possible to be performed and the relevant data are no longer available. Therefore, the Total Number of Participants Affected in Other AEs Table is currently populated with the highest value within the Other AEs table.
Arm/Group | Cervarix Pooled Group | Engerix-B Pooled Group
All-Cause Mortality (participants affected / at risk) | 0/14837 | 0/17338
Serious Adverse Events (participants affected / at risk) | 188/14837 | 152/17338
Other Adverse Events (participants affected / at risk) | 506/643 | 411/1047
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervarix Pooled Group (N=14837) | Engerix-B Pooled Group (N=17338)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 12 (12) | 14 (14)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 7 (7) | 15 (15)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 5 (5) | 3 (3)
Appendicitis perforated (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Genital infection (Infections and infestations) | 0 (0) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 4 (4) | 1 (1)
Muscle abscess (Infections and infestations) | 1 (1) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 4 (4) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic renal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 13 (13) | 25 (25)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Astrocytoma, low grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Cataplexy (Nervous system disorders) | 2 (2) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 2 (2)
Guillain-barre syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 2 (2) | 1 (1)
Narcolepsy (Nervous system disorders) | 2 (2) | 1 (1)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 10 (10) | 15 (15)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 32 (32) | 18 (20)
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 2 (3)
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 10 (11) | 3 (3)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 5 (5)
Peripartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 11 (11) | 6 (6)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Disturbance in social behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Emotional disorder of childhood (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Hypnagogic hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Panic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep attacks (Psychiatric disorders) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis and uveitis syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Testicular torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Henoch-schonlein purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Behcet's syndrome (Vascular disorders) | 0 (0) | 1 (1)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Basedow's disease (Endocrine disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cervarix Pooled Group (N=643) | Engerix-B Pooled Group (N=1047)
Pain (General disorders) | 506/603 | 251/1028 — Solicited symptom during the 7-day post-vaccination period (across doses).
Redness (General disorders) | 169/603 | 131/1028 — Solicited symptom during the 7-day post-vaccination period (across doses).
Arthralgia (General disorders) | 107/604 | 97/1028 — Solicited symptom during the 7-day post-vaccination period (across doses).
Fatigue (General disorders) | 291/604 | 411/1028 — Solicited symptom during the 7-day post-vaccination period (across doses).
Fever (Axillary) (General disorders) | 48/604 | 85/1028 — Solicited symptom during the 7-day post-vaccination period (across doses).
Gastrointestinal (General disorders) | 106/604 | 163/1028 — Solicited symptom during the 7-day post-vaccination period (across doses).
Headache (General disorders) | 261/604 | 371/1028 — Solicited symptom during the 7-day post-vaccination period (across doses).
Nasopharyngitis (Infections and infestations) | 33 | 17 — Unsolicited symptom during the 30-day post-vaccination period (across doses).
Swelling (General disorders) | 131/603 | 46/1028 — Solicited symptom during the 7-day post-vaccination period (across doses).
Myalgia (General disorders) | 321/604 | 250/1028 — Solicited symptom during the 7-day post-vaccination period (across doses).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.